CLINICAL TRIAL: NCT01238614
Title: Universal Screening for Maternal Depression With the CHICA System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Paul Biondich, IUPUI
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: MLM-CHICA-K-MD; K22LM009160 (NIH)
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2010-11

CONDITIONS: Maternal Depression
Keywords: maternal depression; clinical decision support

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PSF-JIT (Experimental): Mothers in this arm receive prescreening questions and clinicians receive just-in-time handouts to aid in diagnosis.
  Interventions: Other: CHICA PSF plus JIT
- PSF (Experimental): Mothers in this arm receive screening questions on the prescreener form
  Interventions: Other: CHICA maternal depression PSF
- Control (Placebo Comparator): Mothers in this arm receive no maternal depression CHICA additional care
  Interventions: Other: Control

INTERVENTIONS:
Other: CHICA PSF plus JIT
  Arms: PSF-JIT
Other: CHICA maternal depression PSF
  Arms: PSF
Other: Control
  Arms: Control

SUMMARY:
The CHICA system is a clinical decision support system that uses adaptive turnaround documents to provide point-of-care information to clinicians. We will be studying whether it can help in the diagnosis and referral of mothers with maternal depression.

ELIGIBILITY:
Inclusion Criteria:

* All families of patients age 0 to 15 months

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3250 (Actual)
Dates: Start 2007-10; Primary Completion 2009-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Percent of mothers screening positive for maternal depression. | 1 year after child's birth

SECONDARY OUTCOMES:
Percent of mothers diagnosed with maternal depression | one year after child's birth

CONTACTS AND LOCATIONS:
Locations (1):
- CHSR, Indianapolis, Indiana, United States